CLINICAL TRIAL: NCT00926289
Title: A Randomised, Double-blind, Double Dummy, Active Controlled, Parallel Group, Forced Titration Study to Compare the Fixed-dose Combination of Telmisartan 80mg Plus Hydrochlorothiazide 25mg (T80/HCTZ25) Versus Telmisartan 80mg (T80) Monotherapy as First Line Therapy in Patients With Grade 2 or Grade 3 Hypertension (Systolic Blood Pressure (SBP) >=160 mmHg and Diastolic Blood Pressure (DBP) >=100 mmHg)
Brief Title: Telmisartan 80mg Plus Hydrochlorothiazide 25mg First Line in Moderate or Severe Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.550; 2008-007711-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

ARMS (2):
- Telmisartan (Active Comparator): Telmisartan 80 mg
  Interventions: Drug: Telmisartan
- Telmisartan/hydrochlorothiazide (Experimental): Telmisartan80mg/Hydrochlorothiazide25mg
  Interventions: Drug: Telmisartan; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan — Telmisartan 80mg
  Arms: Telmisartan
Drug: Telmisartan — Telmisartan 80mg
  Arms: Telmisartan/hydrochlorothiazide
Drug: Hydrochlorothiazide — Hydrochlorothiazide25mg
  Arms: Telmisartan/hydrochlorothiazide

SUMMARY:
The primary objective of this trial is to demonstrate that the fixed-dose combination of T80/HCTZ25 is superior as first line therapy in reducing seated trough cuff Systolic Blood Pressure(SBP) compared to the monotherapy of T80 in patients with grade 2 or grade 3 hypertension (SBP>=160 mmHg and Diastolic Blood Pressure(DBP)>=100 mmHg).

ELIGIBILITY:
Inclusion criteria:

1. Ability to provide written informed consent in accordance with Good Clinical Practice and local legislation;
2. Age 18 years or older;
3. Patients with grade 2 or grade 3 hypertension as defined SBP>=160 mmHg and DBP>=100 mmHg at randomization
4. Ability to stop any current antihypertensive therapy without unacceptable risk to the patient (Investigator's discretion)

Exclusion criteria:

1. Pre-menopausal women (last menstruation <=1 year prior to signing informed consent) who: a) are not surgically sterile; or b) are nursing, or c) are pregnant, or d) are of childbearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the trial. The only acceptable methods of birth control are: Intra-Uterine Device (IUD), Oral contraceptives, Implantable or injectable contraceptives, Estrogen patch Hormonal birth control should have been in use for at least three months before the study and continue at least until the next menstrual period after completing the study.
2. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 a.m.
3. Known or suspected secondary hypertension (e.g., renal artery stenosis orphaeochromocytoma)
4. Mean in-clinic seated cuff SBP>= 200 mmHg and/or DBP >=120 mmHg
5. Renal dysfunction as defined by the following laboratory parameters: Serum creatinine >3.0 mg/dL (or >265 umol/L) and/or known creatinine clearance of <30 ml/min and/or clinical markers of severe renal impairment.
6. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney
7. Clinically relevant hypokalemia or hyperkalemia (i.e., <3.5 mmol/L or >5.5 mmol/L, may be rechecked for suspected error in result)
8. Uncorrected sodium or volume depletion
9. Primary aldosteronism.
10. Hereditary fructose intolerance
11. Biliary obstructive disorders (e.g., cholestasis) or hepatic insufficiency
12. Congestive heart failure New York Heart Association functional class Congestive Heart Failure III-IV (Refer to Appendix 10.3)
13. Contra-indication to a placebo run-in period (e.g., stroke with-in the past 6 months, myocardial infarction, cardiac surgery, percutaneous transluminal coronary angioplasty, unstable angina or coronary artery bypass graft within the past 3 months prior to start of run in period)
14. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the Investigator
15. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
16. Patients whose diabetes has not been stable and controlled for at least the past 3 months as defined by an Glycosylated Hemoglobin >=10%
17. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin-II receptor antagonists
18. History of drug or alcohol dependency within 6 months prior to signing the informed consent form
19. Concomitant administration of any medications known to affect blood pressure, except medications allowed by the protocol
20. Any investigational drug therapy within 1 month of signing the informed consent
21. Known hypersensitivity to any component of the trial drugs (telmisartan, hydrochlorothiazide, or placebo)
22. History of non-compliance or inability to comply with prescribed medications or protocol procedures (less than 80% or more than 120%, especially during run-in)
23. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (106):
- United States (18):
  - 502.550.01008 Boehringer Ingelheim Investigational Site, Athens, Alabama
  - 502.550.01019 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 502.550.01015 Boehringer Ingelheim Investigational Site, Lomita, California
  - 502.550.01003 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 502.550.01014 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 502.550.01002 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 502.550.01011 Boehringer Ingelheim Investigational Site, New Iberia, Louisiana
  - 502.550.01009 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 502.550.01018 Boehringer Ingelheim Investigational Site, Olive Branch, Mississippi
  - 502.550.01006 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 502.550.01016 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 502.550.01007 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 502.550.01005 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 502.550.01001 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 502.550.01017 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 502.550.01020 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 502.550.01012 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 502.550.01004 Boehringer Ingelheim Investigational Site, Arlington, Virginia
- Bulgaria (10):
  - 502.550.35901 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35902 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35905 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35908 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35909 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35910 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35911 Boehringer Ingelheim Investigational Site, Sofia
  - 502.550.35906 Boehringer Ingelheim Investigational Site, Stara Zagora
- China (8):
  - 502.550.86004 Boehringer Ingelheim Investigational Site, Changsha
  - 502.550.86003 Boehringer Ingelheim Investigational Site, Guangzhou, Guangdong Province
  - 502.550.86008 Boehringer Ingelheim Investigational Site, Qingdao
  - 502.550.86001 Boehringer Ingelheim Investigational Site, Shanghai
  - 502.550.86002 Boehringer Ingelheim Investigational Site, Shanghai
  - 502.550.86009 Boehringer Ingelheim Investigational Site, Shenyang
  - 502.550.86007 Boehringer Ingelheim Investigational Site, Tianjin
  - 502.550.86010 Boehringer Ingelheim Investigational Site, Zhengzhou
- France (28):
  - 502.550.3302D Boehringer Ingelheim Investigational Site, Aigrefeuille S/Maine
  - 502.550.3305I Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 502.550.3305G Boehringer Ingelheim Investigational Site, Aubagne
  - 502.550.3301H Boehringer Ingelheim Investigational Site, Briollay
  - 502.550.3301K Boehringer Ingelheim Investigational Site, Cholet
  - 502.550.3302I Boehringer Ingelheim Investigational Site, Corsept
  - 502.550.3302C Boehringer Ingelheim Investigational Site, Donges
  - 502.550.3302B Boehringer Ingelheim Investigational Site, La Montagne
  - 502.550.3306A Boehringer Ingelheim Investigational Site, Louvigné-de-Bais
  - 502.550.3303A Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3303D Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3303F Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3304A Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3304D Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3304F Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3304J Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3305A Boehringer Ingelheim Investigational Site, Marseille
  - 502.550.3301A Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 502.550.3301I Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 502.550.3302A Boehringer Ingelheim Investigational Site, Nantes
  - 502.550.3302E Boehringer Ingelheim Investigational Site, Nantes
  - 502.550.3301E Boehringer Ingelheim Investigational Site, Parçay-les-Pins
  - 502.550.3303C Boehringer Ingelheim Investigational Site, Roquevaire
  - 502.550.3302G Boehringer Ingelheim Investigational Site, Saint Aubin Les Châteaux
  - 502.550.3306F Boehringer Ingelheim Investigational Site, Saint-Jouan-des-Guérets
  - 502.550.3301F Boehringer Ingelheim Investigational Site, Segré
  - 502.550.3307A Boehringer Ingelheim Investigational Site, Thouars
  - 502.550.3301J Boehringer Ingelheim Investigational Site, Vihiers
- Georgia (8):
  - 502.550.99501 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99502 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99503 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99504 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99505 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99506 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99507 Boehringer Ingelheim Investigational Site, Tbilisi
  - 502.550.99508 Boehringer Ingelheim Investigational Site, Tbilisi
- Romania (11):
  - 502.550.40002 Boehringer Ingelheim Investigational Site, Baia Mare Maramures
  - 502.550.40003 Boehringer Ingelheim Investigational Site, Brăila
  - 502.550.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 502.550.40010 Boehringer Ingelheim Investigational Site, Bucharest
  - 502.550.40012 Boehringer Ingelheim Investigational Site, Bucharest
  - 502.550.40009 Boehringer Ingelheim Investigational Site, Cluj-Napoca
  - 502.550.40011 Boehringer Ingelheim Investigational Site, Cluj-Napoca
  - 502.550.40006 Boehringer Ingelheim Investigational Site, Iași
  - 502.550.40004 Boehringer Ingelheim Investigational Site, Oradea
  - 502.550.40005 Boehringer Ingelheim Investigational Site, Sibiu
  - 502.550.40008 Boehringer Ingelheim Investigational Site, Tg. Mures
- Russia (10):
  - 502.550.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 502.550.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 502.550.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 502.550.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 502.550.07005 Boehringer Ingelheim Investigational Site, Moscow
  - 502.550.07006 Boehringer Ingelheim Investigational Site, Moscow
  - 502.550.07007 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 502.550.07008 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 502.550.07009 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 502.550.07010 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Korea (13):
  - 502.550.82008 Boehringer Ingelheim Investigational Site, Cheonan
  - 502.550.82009 Boehringer Ingelheim Investigational Site, Daegu
  - 502.550.82001 Boehringer Ingelheim Investigational Site, Goyang
  - 502.550.82003 Boehringer Ingelheim Investigational Site, Gwangju
  - 502.550.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82011 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82012 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82013 Boehringer Ingelheim Investigational Site, Seoul
  - 502.550.82004 Boehringer Ingelheim Investigational Site, Suwon
  - 502.550.82010 Boehringer Ingelheim Investigational Site, Wŏnju

REFERENCES:
- [Derived] Zhu DL, Bays H, Gao P, Mattheus M, Voelker B, Ruilope LM. Efficacy and tolerability of initial therapy with single-pill combination telmisartan/hydrochlorothiazide 80/25 mg in patients with grade 2 or 3 hypertension: a multinational, randomized, double-blind, active-controlled trial. Clin Ther. 2012 Jul;34(7):1613-24. doi: 10.1016/j.clinthera.2012.05.007. Epub 2012 Jun 19. PMID 22717420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 894 patients were entered (randomised) into the study; however, of these, 6 were not treated. Therefore 888 patients actually entered into treatment.
Groups:
- Telmisartan 40/80 mg: Telmisartan 40mg once daily for 1 week with forced titration to 80 mg for 6 weeks
- Telmisartan 40/80 mg + HCTZ (Hydrochlorothiazide) 12.5/25 mg: fixed combination of Telmisartan 40mg and HCTZ 12.5 mg once daily for 1 week with forced titration to T80+HCTZ25 for 6 weeks
Period: Overall Study
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ (Hydrochlorothiazide) 12.5/25 mg
Started | 294 (Number of treated patients) | 594 (Number of treated patients)
Completed | 269 | 558
Not Completed | 25 | 36
Not completed — Adverse Event | 9 | 11
Not completed — Protocol Violation | 8 | 12
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Telmisartan 40/80 mg + HCTZ 12.5/25 mg: fixed combination of Telmisartan 40mg and HCTZ 12.5 mg once daily for 1 week with forced titration to T80+HCTZ25 for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg | Total
Number analyzed (Participants) | 294 | 594 | 888
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (11.9) | 56.8 (11.3) | 57.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 285 | 410
  Male | 169 | 309 | 478

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated Trough Cuff Systolic Blood Pressure (SBP) to Week 7
Description: The SBP value at baseline was subtracted from the SBP value at Week 7.
Time Frame: Baseline and Week 7
Population: The Full Analysis Set (FAS) included all patients in the treated set who provide a baseline trough cuff BP measurement and at least one seated trough cuff BP measurement following titration to target therapy (T80+H25 or T80), taken on the same arm
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 263 | 541
mmHg | -28.5 (0.88) | -37.0 (0.62)
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; Fixed effects of treatment, week, treatment-by-week interaction, country with the continuous covariates of baseline and baseline-by-week interaction; Mean Difference (Final Values) = -8.5, 95% CI [-10.6 to -6.4]

2. Secondary Outcome: Change From Baseline in Mean Seated Trough Cuff SBP to Week 5
Description: The SBP value at baseline was subtracted from the SBP value at Week 5.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 270 | 550
mmHg | -28.6 (0.86) | -35.8 (0.61)
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.3, 95% CI [-9.3 to -5.2]

3. Secondary Outcome: Change From Baseline in Mean Seated Trough Cuff SBP to Week 3
Description: The SBP value at baseline was subtracted from the SBP value at Week 3.
Time Frame: Baseline and Week 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 276 | 567
mmHg | -26.5 (0.87) | -33.3 (0.61)
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.8, 95% CI [-8.8 to -4.7]

4. Secondary Outcome: Change From Baseline in Mean Seated Trough Cuff Diastolic Blood Pressure (DBP) to Week 7
Description: The DBP value at baseline was subtracted from the DBP value at Week 7.
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 263 | 541
mmHg | -15.4 (0.55) | -18.6 (0.38)
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.2, 95% CI [-4.5 to -1.9]

5. Secondary Outcome: Number of Patients With SBP Control (SBP < 140 mmHg) at Week 7
Description: SBP control is defined as SBP < 140 mmHg.
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants | 122 | 363
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.36, 95% CI [1.74 to 3.21]

6. Secondary Outcome: Number of Patients With SBP Control (SBP < 140 mmHg) at Week 5
Description: SBP control is defined as SBP < 140 mmHg
Time Frame: Week 5 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 284 | 572
Participants | 119 | 355
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.30, 95% CI [1.70 to 3.12]

7. Secondary Outcome: Number of Patients With SBP Control (SBP < 140 mmHg) at Week 3
Description: SBP control is defined as SBP < 140 mmHg
Time Frame: Week 3 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 276 | 567
Participants | 97 | 306
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.19, 95% CI [1.60 to 3.01]

8. Secondary Outcome: Number of Patients With DBP Control (DBP < 90 mmHg) at Week 7
Description: DBP control is defined as DBP<90 mmHg
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants | 150 | 389
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.00, 95% CI [1.46 to 2.73]

9. Secondary Outcome: Number of Patients With DBP Control (DBP < 90 mmHg) at Week 5
Description: DBP control is defined as DBP<90 mmHg
Time Frame: Week 5 timepoint
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 284 | 572
participants | 150 | 391
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.02, 95% CI [1.48 to 2.76]

10. Secondary Outcome: Number of Patients With DBP Control (DBP < 90 mmHg) at Week 3
Description: DBP control is defined as DBP<90 mmHg
Time Frame: Week 3 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 276 | 567
Participants | 131 | 343
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Adjustment for continuous covariate of baseline and fixed effect country; Odds Ratio (OR) = 1.74, 95% CI [1.28 to 2.37]

11. Secondary Outcome: Number of Patients With Blood Pressure (BP) Control at Week 7
Description: BP control is defined as SBP<140 mmHg and DBP < 90 mmHg and is adjusted for baseline SBP
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants | 99 | 318
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline (SBP), treatment and country as fixed effects; Odds Ratio (OR) = 2.39, 95% CI [1.76 to 3.26]

12. Secondary Outcome: Number of Patients With BP Control at Week 7
Description: BP control is defined as SBP<140 mmHg and DBP < 90 mmHg and is adjusted for baseline DBP
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants | 99 | 318
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline (DBP), treatment and country as fixed effects; Odds Ratio (OR) = 2.42, 95% CI [1.78 to 3.29]

13. Secondary Outcome: Number of Patients With Systolic Blood Pressure (SBP) Response at Week 7
Description: SBP response is defined as SBP<140 mmHg or a reduction of >= 15 mmHg
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants | 233 | 527
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.62, 95% CI [1.70 to 4.04]

14. Secondary Outcome: Number of Participants With DBP Response at Week 7
Description: DBP response is defined as DBP<90 mmHg or a reduction of >= 10 mmHg
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants | 202 | 483
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for continuous covariate of baseline, treatment and country as fixed effects; Odds Ratio (OR) = 2.23, 95% CI [1.57 to 3.16]

15. Secondary Outcome: BP Categories at Week 7
Description: BP categories comprise:
  * BP optimal (SBP <120 mmHg and DBP <80 mmHg)
  * BP normal (SBP <130 mmHg and DBP <85 mmHg but not 'optimal')
  * BP high normal (SBP <140 mmHg and DBP <90 mmHg but not 'normal')
  * Grade 1 hypertension (SBP <160 mmHg and DBP <100 mmHg but not 'high normal')
  * Grade 2 hypertension (SBP <180 mmHg and DBP <110 mmHg but not 'Grade 1 hypertension')
  * Grade 3 hypertension (SBP ≥180 mmHg or DBP ≥110 mmHg)
Time Frame: Week 7 timepoint
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Number analyzed (Participants) | 285 | 573
Participants
  BP optimal | 6 | 44
  BP normal | 36 | 136
  BP high normal | 57 | 138
  Grade 1 hypertension | 120 | 186
  Grade 2 hypertension | 44 | 58
  Grade 3 hypertension | 22 | 11
Statistical Analysis 1: Comparison: Telmisartan 40/80 mg vs Telmisartan 40/80 mg + HCTZ 12.5/25 mg; T80+HCTZ25 versus T80 monotherapy; Test type: Superiority or Other; p < 0.0001, Van Elteren test stratified for country

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Telmisartan 40/80 mg | Telmisartan 40/80 mg + HCTZ 12.5/25 mg
Serious Adverse Events (participants affected / at risk) | 1/294 | 0/594
Other Adverse Events (participants affected / at risk) | 0/294 | 0/594
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40/80 mg (N=294) | Telmisartan 40/80 mg + HCTZ 12.5/25 mg (N=594)
Epilepsy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.